CLINICAL TRIAL: NCT02696980
Title: Increased Lung Volume as Rescue Therapy for Asthma
Brief Title: PEEP as Rescue Therapy for Asthmatics With Elevated BMI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Anne Dixon, Professor of Medicine, University of Vermont
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: M16-060
Record Dates: First submitted 2016-02-23; First posted 2016-03-02 (Estimated); Results first posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-06

CONDITIONS: Asthma
Keywords: obesity; asthma
MeSH Terms: conditions — Asthma; Obesity | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Rescue (Experimental): Intervention: Positive expiratory pressure (PEEP) 10 will be applied after the administration of methacholine
  Interventions: Device: Positive Expiratory Pressure
- Prophylaxis (Experimental): Intervention: Positive expiratory pressure (PEEP) 10 will be applied during the administration of methacholine
  Interventions: Device: Positive Expiratory Pressure
- No PEEP (Placebo Comparator): Intervention: Positive expiratory pressure (PEEP) 0 will be applied during the administration of methacholine
  Interventions: Device: Positive Expiratory Pressure

INTERVENTIONS:
Device: Positive Expiratory Pressure — Patient will exhale against positive expiratory pressure 0 mm or 10 mm while inhaling methacholine
  Other Names: PEEP

SUMMARY:
The purpose of this study is to test the effect of increasing lung volume with a simple hand-held device to both prevent, and also to relieve, airway constriction in people with asthma and a BMI ≥ 30 kg/m2.

Twenty people with late onset non-allergic asthma and a BMI of ≥ 30 kg/m2 will be recruited. The efficacy of elevating lung volume on both preventing and reversing bronchoconstriction will be tested. Lung volume will be modulated by breathing out against a small level of resistance (positive expiratory pressure).

DETAILED DESCRIPTION:
This study will investigate whether PEEP can prevent and/or reverse bronchoconstriction in asthmatics with a BMI > 30 kg/m2.

People with late-onset non-allergic asthma that develops in the setting of obesity do not respond well to conventional asthma medications, likely because all treatments for asthma have been developed to treat early-onset allergic disease in lean patients. There is a critical need to understand the pathophysiology of airway disease in late-onset, non-allergic obese asthmatics, in order to develop therapies to target this disease.

Airway hyperresponsiveness (AHR) is a defining characteristic in asthma. Lung function tests in individuals with late onset asthma in the setting of obesity are suggestive of distal airway closure rather than airway narrowing as a cause of hyperresponsiveness; these individuals tend to have more collapsible lung peripheries than obese individuals who do not develop asthma. If late onset asthma in obesity is related to a tendency of airways to close, it should respond to therapies designed to keep airways open, such as Positive End-Expiratory Pressure (PEEP).

The purpose of this study is to investigate the efficacy of PEEP on prevention and reversal of bronchoconstriction in obese people with asthma. This will be achieved by investigating the efficacy of PEEP therapy on preventing and reversing bronchoconstriction in response to the inhalation of methacholine, while measuring changes in respiratory impedance using the forced oscillation method.

Participants will initially perform a conventional methacholine challenge test.

Participants will return for 2 visits in which methacholine will be administered concurrently with varying levels of PEEP (using PEEP to prevent bronchoconstriction) while measuring changes in respiratory impedance using the forced oscillation method.

Participants will return for another 2 visits in which PEEP will be administered subsequent to methacholine challenge (using PEEP to reverse bronchoconstriction) while measuring changes in respiratory impedance using the forced oscillation method.

These studies will be completed over 5 visits.

ELIGIBILITY:
Inclusion Criteria:

* PC20 to methacholine < 16 mg/ml
* Asthma diagnosis when ≥ 18 years of age
* Serum Immunoglobulin E < 100 IU/ml
* Ages ≥ 18 years
* BMI ≥ 30 kg/m2

Exclusion Criteria:

* Asthma exacerbation (defined as a hospitalization, ED visit, urgent care visit for asthma or new corticosteroids for asthma) in prior 6 weeks.
* Forced Expiratory Volume in 1 second < 60 % predicted
* Other significant disease that in the opinion of the investigator would interfere with study
* Inability to perform required testing.
* Smoking within last 6 months.
* ≥ 20 pack year smoking history
* Inability to provide informed consent
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-04; Primary Completion 2019-04 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Dixon, BM BCh, Principal Investigator — University of Vermont
Locations (1):
- Vermont Lung Center, Colchester, Vermont, United States

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in the archival literature, and this will include a complete description of experimental and analytical methods used. All original experimental data will be stored and available to interested investigators with appropriate regulatory approvals in place.
Supporting Information: CSR
Time Frame: Clinical study report published December 2021.
URL: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8714981/

REFERENCES:
- [Background] Al-Alwan A, Bates JH, Chapman DG, Kaminsky DA, DeSarno MJ, Irvin CG, Dixon AE. The nonallergic asthma of obesity. A matter of distal lung compliance. Am J Respir Crit Care Med. 2014 Jun 15;189(12):1494-502. doi: 10.1164/rccm.201401-0178OC. PMID 24821412
- [Background] Chapman DG, Irvin CG, Kaminsky DA, Forgione PM, Bates JH, Dixon AE. Influence of distinct asthma phenotypes on lung function following weight loss in the obese. Respirology. 2014 Nov;19(8):1170-7. doi: 10.1111/resp.12368. Epub 2014 Aug 19. PMID 25138203

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between 2016-2019. There was a minor delay to the enrollment timeline relative to the proposed starting date due to staffing changes. The uploaded protocol is an IRB approved document. Given that the study is now complete, the IRB record has been closed out and further modification of this protocol is not possible.
Groups:
- All Patients: Cross over study: Intervention:
  1. Positive expiratory pressure (PEP) 10 applied for 2.5 minutes after administration of participant's PC20 dose of methacholine (dose producing a 20% fall in FEV1).
  2. PEP 10 during and after for 2.5 minutes after participant's PC20 dose of methacholine
  3. PEP 0 during and for 2.5 minutes after administration of participant's PC20 dose of methacholine
  All participants were studied in conditions 1, 2 and 3 on separate days, order of visits were randomized
Period: Overall Study
Arm/Group | All Patients
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants Assigned to Intervention in Cross Over Design: participants underwent the following studies and intervention
  1. PEP 10 after methacholine 3. PEP 10 during methacholine 3. PEP 0
Arm/Group | All Study Participants Assigned to Intervention in Cross Over Design
Number analyzed (Participants) | 18
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52 [40 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Central and Peripheral Elastance
Description: Investigators compare changes in respiratory system elastance to methacholine. Respiratory system impedance was measured at the 8-min time point and fit with the two-compartment series model of respiratory mechanics. The elastances of the central and distal compartments obtained from good quality fits of this model are reported for each of the following conditions:
  V2: PEP of 0 was administered during (0-4.5 min) and after (4.5-8 min) methacholine administration.
  V3: PEP of 0 was administered during (0-4.5 min) and PEP of 10 cmH2O after (4.5-8 min) methacholine administration.
  V4: This is a repeat of V2 above to test for stability of the response. V5: PEP of 10 cmH2O was administered both during (0-4.5 min) and after (4.5-8 min) methacholine administration.
  V1 was a baseline visit to establish physiologic parameters required for conducting Visits 2-5. There are no outcome measures for Visit 1.
Time Frame: The end of the experiment (at the 8-min time point)
Measure: Mean (Standard Error); unit: cmH2O/L
Groups:
- Visit 2; Visit 4: PEP 0 during and after methacholine
- Visit 3: PEP 0 during methacholine, PEP 10 cmH2O after methacholine
- Visit 5: PEP 10 cmH2O during and after methacholine
Arm/Group | Visit 2 | Visit 3 | Visit 4 | Visit 5
Number analyzed (Participants) | 10 | 10 | 13 | 10
cmH2O/L
  Central Elastance | 391 (86) | 461 (82) | 587 (299) | 334 (60)
  Peripheral Elastance | 103 (50) | 82 (16) | 162 (33) | 42 (16)

ADVERSE EVENTS:
Time Frame: Duration of each study visit (during methacholine, and for 30 minutes after)
Description: reported by patient to research coordinator
Groups:
- Rescue: Cross over study: Intervention: Positive expiratory pressure (PEP) 10 will be applied after the administration of methacholine, during administration and after methacholine, and PEP 0 during and after metacholine at separate visits
Arm/Group | Rescue
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-05): https://cdn.clinicaltrials.gov/large-docs/80/NCT02696980/Prot_SAP_001.pdf
  • Informed Consent Form (2018-03-05): https://cdn.clinicaltrials.gov/large-docs/80/NCT02696980/ICF_000.pdf